CLINICAL TRIAL: NCT05546359
Title: Randomized, Double-blind, Phase 2/3 Study of IV Amisulpride as Prevention of Post-operative Nausea and Vomiting in Pediatric Patients
Brief Title: Study of Intravenous Amisulpride for Prophylaxis of Post-operative Nausea and Vomiting (PONV) in Pediatric Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Acacia Pharma Ltd (Industry)
Collaborators: Amicus CD LLC (Unknown); Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DP10027
Record Dates: First submitted 2022-09-12; First posted 2022-09-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Nausea and Vomiting, Postoperative
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Amisulpride; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stage 1 - Group 1: IV amisulpride 0.035 mg/kg + IV dexamethasone (Experimental): Stage 1 - Group 1: IV amisulpride 0.035 mg/kg + IV dexamethasone
  Interventions: Drug: Amisulpride Injection; Drug: Dexamethasone
- Stage 1 - Group 2: IV amisulpride 0.07 mg/kg + IV dexamethasone (Experimental): Stage 1 - Group 2: IV amisulpride 0.07 mg/kg + IV dexamethasone
  Interventions: Drug: Amisulpride Injection; Drug: Dexamethasone

INTERVENTIONS:
Drug: Amisulpride Injection — Dose finding treatment for continuation to phase 3
  Other Names: Barhemsys
Drug: Dexamethasone — Standard of care treatment
  Other Names: Decadron

SUMMARY:
Randomized, double-blind, pediatric trial of amisulpride for prophylaxis of post operative nausea and vomiting

DETAILED DESCRIPTION:
Randomized, double-blind, Phase 2/3 study of IV amisulpride as prevention of post-operative nausea and vomiting in pediatric patients

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged from full-term birth to 17 years of age
2. Signed informed consent form and/or assent and willingness of patient and parents to participate in the trial
3. Patients undergoing non-emergency surgery, preferentially eye surgery, adenotonsillectomy or otoplasty, under general anesthesia (other than total intravenous anesthesia with propofol) expected to last at least 30 minutes from induction of anesthesia to removal of Endotracheal tube (ETT) or Laryngeal mask airway (LMA)
4. American Society of Anesthesiologists (ASA) risk score I-III
5. For females of child-bearing potential: ability and willingness to use a highly effective form of contraception (as defined in ICH M3 guidance, e.g., true (not periodic) abstinence from sexual intercourse, surgical sterilization (of subject or partner), combined oral contraceptive pill, or any other method or combination of methods with a failure rate generally considered to be <1% per year) between the date of screening and at least 48 hours after administration of study drug.

Exclusion Criteria:

1. Patients scheduled to undergo transplant or Central Nervous System (CNS) surgery
2. Patients scheduled to receive only a local anesthetic and/or regional neuraxial (intrathecal or epidural) block (without general anesthesia) or to receive general anesthesia involving total intravenous anesthesia (TIVA) with propofol
3. Patients who, in the opinion of the Investigator, are expected to remain ventilated for a significant period after surgery
4. Patients who are expected to need a naso- or orogastric tube in situ after surgery is completed
5. Patients who are expected to receive systemic pre/peri-operative corticosteroid therapy other than as anti-emetic prophylaxis
6. Patients receiving amisulpride for any indication within the 2 weeks prior to randomization
7. Patients known to be allergic to amisulpride or any of the excipients of amisulpride drug product; or to dexamethasone or ondansetron
8. Patients with a significant ongoing history of vestibular disease or dizziness
9. Patients being treated with regular anti-emetic therapy (dosed at least three times per week), which is still ongoing less than 1 week prior to screening
10. Patients being treated with levodopa, or any other dopamine D2-agonist
11. Patients who are pregnant or breast feeding
12. Patients with congenital long QT interval (QT) syndrome
13. Patients with a tumor of the anterior pituitary
14. Patients who have received emetogenic anti-cancer chemotherapy in the previous 4 weeks
15. Any other concurrent disease or illness that, in the opinion of the investigator makes the patient unsuitable for the study
16. Patients who have previously participated in this study or who have participated in another interventional clinical study involving pharmacological therapy within the previous 28 days (or longer exclusion period, if required by national or local regulations)
17. Where local laws/regulations require: patients under legal protection

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 453 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Evaluate Complete Response | 1 Day
  Defined as no vomiting/retching (absence of PONV) and no use of anti-emetic rescue medication, during the first 24 hours after completion of surgery. Subjects will be questioned and assessed.

SECONDARY OUTCOMES:
Occurrence of post-operative vomiting/retching | 1 Day
  Subjects considered able to understand and provide a meaningful response should be asked if they have nausea ("feel sick" or other equivalent words) at the following times after completion of surgery (wound closure), unless an episode of PONV or discharge of the subject from the site has already occurred prior to the time point: 1 hour, 2 hours, 6 hours and 24 hours or when they first vomit, retch or receive rescue medication. In subjects aged ≥ 6 years, at the above time points and for any spontaneously reported nausea episode, nausea severity should be scored using the validated 6-point Baxter Retching Faces (BARF) scale.
Use of rescue medication | 1 Day
  Document use of rescue medication.
Occurrence and severity of post-operative nausea | 1 Day
  An episode of nausea should be recorded any time that a subject spontaneously complains of nausea (including a request for rescue medication due to nausea). Subjects considered able to understand and provide a meaningful response should be asked if they have nausea ("feel sick" or other equivalent words) at the following times after completion of surgery (wound closure), unless an episode of PONV or discharge of the subject from the site has already occurred prior to the time point: 1 hour, 2 hours, 6 hours and 24 hours or when they first vomit, retch or receive rescue medication. In subjects aged ≥ 6 years, at the above time points and for any spontaneously reported nausea episode, nausea severity should be scored using the validated 6-point Baxter Retching Faces (BARF) scale.
Time to emergence of PONV | 1 Day
  Observe for, question and document emergence of vomiting/retching and nausea. In subjects aged ≥ 6 years, at specified time points and for any spontaneously reported nausea episode, nausea severity should be scored using the validated 6-point Baxter Retching Faces (BARF) scale.
Time to emergence of vomiting/retching, significant nausea, and rescue medication, individually | 1 Day
  Observe for emergence of vomiting/retching, determine significance of nausea, and note rescue medication, individually.
Different variables during different time ranges after the end of surgery (0-2 h, 2-6 h and 6-24 h) | 1 Day
  Subjects considered able to understand and provide a meaningful response should be asked if they have nausea ("feel sick" or other equivalent words) at the following times after completion of surgery (wound closure), unless an episode of PONV or discharge of the subject from the site has already occurred prior to the time point: 1 hour, 2 hours, 6 hours and 24 hours or when they first vomit, retch or receive rescue medication. In subjects aged ≥ 6 years, at the above time points and for any spontaneously reported nausea episode, nausea severity should be scored using the validated 6-point Baxter Retching Faces (BARF) scale.
The above variables in the sub-groups of patients who did and did not receive opioid analgesia | 1 Day
  Concomitant medications will be reviewed.
Safety: The nature and frequency of adverse events and laboratory and electrocardiography (ECG) abnormalities | 7 Days
  Adverse events, laboratory and ECG abnormalities will be noted. Blood samples should be drawn at screening (unless recent pre-existing results are available) and again post-operatively, as soon as practically possible after the patient's entry to the post-anesthesia care unit, recovery room or equivalent, and in any event within 1 hour after the end of surgery. Twelve-lead ECGs will be collected at screening. An ECG already taken as part of medical care within the period of 2 weeks prior to screening may be used to determine eligibility and to provide baseline ECG data.
  In the peri-/post-operative period, continuous Holter monitoring of the ECG will be performed, from at least 10 minutes prior until at least 2 hours after the start of administration of amisulpride study medication.
Key pharmacokinetics parameter - Peak Plasma Concentration | 1 Day
  Plasma samples will be drawn as required at specified timepoints to determine the PK profile of peak plasma concentration of amisulpride in subjects.
Key pharmacokinetics parameter - Total Exposure | 1 Day
  Plasma samples will be drawn as required at specified timepoints to determine the PK profile of total exposure of amisulpride in subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Kumar Belani, MD, Principal Investigator — University of Minnesota Masonic Children's Hospital
Locations (14):
- United States (5):
  - Helen Keller Hospital, Sheffield, Alabama
  - Emory Healthcare - Emory University Hospital, Atlanta, Georgia
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Centre - The Montréal Children's Hospital, Montreal, Quebec
- France (2):
  - HCL - Hôpital Mère Enfant, Bron
  - CHU Strasbourg - Hopital Hautepierre, Strasbourg
- Germany (5):
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Ambulantes Operieren Marburg, Marburg, Hesse
  - Universitaetsklinikum Giessen und Marburg GmbH, Marburg, Hesse
  - Universitaetsklinikum Bonn - Klinik für Anaesthesiologie & Operative Intensivmedizin, Bonn, North Rhine-Westphalia
  - Helios Klinikum Aue, Aue

IPD SHARING:
Plan to Share IPD: No